CLINICAL TRIAL: NCT04924985
Title: Goal-Directed Cardiopulmonary Resuscitation in Cardiac Arrest Using a Novel Physiological Target
Brief Title: Goal-directed CPR Using Cerebral Oximetry
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-00354; 1R01HL151732-01 (NIH)
Record Dates: First submitted 2021-06-10; First posted 2021-06-14 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Ischemia; Reperfusion Injury
Keywords: CPR
MeSH Terms: conditions — Ischemia; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiological Feedback CPR (Experimental)
  Interventions: Other: Physiological Feedback CPR
- Non-Physiological (Audiovisual) Feedback CPR (Active Comparator)
  Interventions: Other: Non-Physiological Feedback CPR

INTERVENTIONS:
Other: Non-Physiological Feedback CPR — Non-physiologically guided CPR using AV feedback (integrated into defibrillators)
  Arms: Non-Physiological (Audiovisual) Feedback CPR
Other: Physiological Feedback CPR — Physiological feedback CPR using an optimal regional O2 Saturation (rSO2), End-tidal CO2 (ETCO2) or combined (rSO2/ETCO2) target
  Arms: Physiological Feedback CPR

SUMMARY:
The proposed study is a single-center, randomized controlled pilot trial of adults who suffer in-hospital cardiac arrests. Using cerebral oxygenation and end-tidal carbon dioxide physiological targets to predict survival and neurological outcome, the impact of physiological-feedback CPR will be assessed. 150 adult patients who have a cardiac arrest event at NYU Tisch Hospital will be randomized to one of two treatment groups: (1) Physiological-Feedback CPR or (2) Non-Physiological (Audiovisual) Feedback CPR.

ELIGIBILITY:
Inclusion Criteria:

1. In-hospital cardiac arrest patient
2. Age ≥18 years
3. Age <80 years
4. CPR lasting ≥5 minutes

Exclusion Criteria:

1. Patients < 18 years of age or > 80 years of age
2. Out of hospital cardiac arrest patients
3. ≥3 acute organ failures (defined as acute renal failure requiring dialysis, fulminant liver failure i.e. liver failure with INR≥1.5, respiratory failure requiring mechanical ventilation)
4. Repeat in-hospital cardiac arrest event within 14 days of a prior cardiac arrest
5. Presence of known raised intracranial pressure
6. Presence of known traumatic brain injury or subarachnoid hemorrhage <14 days old, frontal lobe brain tumors or subdural hemorrhage
7. Hyperbilirubinemia >1.0 mg/dl (based on the absorption of near-infrared light by bilirubin)
8. Resuscitation using extra-corporeal membrane oxygenation (ECMO)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Return of Spontaneous Circulation (ROSC) | Day 0

SECONDARY OUTCOMES:
Cerebral Performance Category (CPC) Score | Day 1-2
  Total range of score is 1 (Good cerebral performance) to 5 (Brain death). The higher the score, the worse the clinical condition.
Cerebral Performance Category (CPC) Score | Day 30
  Total range of score is 1 (Good cerebral performance) to 5 (Brain death). The higher the score, the worse the clinical condition.
Change in mean rSO2 during CPR as markers of the quality of resuscitation | Day 0
Change in mean ETCO2 during CPR as markers of the quality of resuscitation | Day 0
Release of interleukin (IL)-6 | Day 0
Release of Lactate | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Sam Parnia, MD, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Sam.Parnia@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT04924985/ICF_000.pdf